CLINICAL TRIAL: NCT04738305
Title: Feasibility and Acceptability of a Dignity Therapy Intervention on Palliative Care Program's Cancer Patients Referring to a Medical Oncology Ward.
Brief Title: Feasibility of Dignity Therapy Intervention on Cancer Patients in Charge to an Hospital Palliative Care Unit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/0007193
Record Dates: First submitted 2021-01-26; First posted 2021-02-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Dignity; Advanced Cancer
Keywords: Hospital palliative care unit
MeSH Terms: interventions — Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dignity Therapy Intervention (Other): All the patients that accepted to participate in the study were provided with Dignity Therapy Intervention. A short-term intervention aimed at reducing existential distress of patients facing with advanced illness.
  Interventions: Other: Dignity Therapy

INTERVENTIONS:
Other: Dignity Therapy — The Italian version Dignity Therapy intervention (Chochinov HM 2015) has been delivered. Intervention questions were not previously delivered to patients.
  DT interview was provided to patients by Specifically trained Nurses. Interviews were audio-recorded and transcribed then revised by the patients to develop the final Generativity Document. Generativity Document was delivered to patients that could share it with their loved ones.

SUMMARY:
Aim of the study was to asses feasibility and acceptability of a nurse delivered Dignity Therapy (DT) intervention on advanced cancer patients referring to an Hospital palliative care unit. To achieve this aim a mixed-method approach using before and after evaluation and semi-structured interviews has been used.

ELIGIBILITY:
Inclusion Criteria:

* advanced cancer patients
* over 3 months life expectancy
* referring to hospital palliative care unit
* performance status (Eastern Cooperative Oncology Group - ECOG) between 0 and 2
* awareness of being affected by an incurable cancer
* cognitive ability to read, understand and fill in a questionnaire in Italian
* willing and able to give written informed consent

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | 1 year
  The number of participants who sign the informed consent form divided by the number who are asked to participate in the study
Retention rate | 1 year
  The number of participants who performed the post intervention assesment divided by the number of enrolled one.
Professionals' experience in implementing DT | 12-18 months
  Semi-structured interviews administered to the three nurses that implemented the higher number of DT interventions. Interview were performed after the last patient completed the post intervention assessment.

SECONDARY OUTCOMES:
Patient dignity-related | Baseline; day 62
  Patient Dignity Inventory (Italian version). Scale range 25-125, higher value means higher dignity-related distress.
Patient feedback | day 62
  The acceptability of Dignity Therapy was assessed by the Italian version of "Dignity Therapy Patient Feedback Questionnaire" survey.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Nunziante, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL - IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chochinov HM. Terapia della dignità: parole per il tempo che rimane. Il pensiero scientifico, 2015.
- [Derived] Nunziante F, Tanzi S, Alquati S, Autelitano C, Bedeschi E, Bertocchi E, Dragani M, Simonazzi D, Turola E, Braglia L, Masini L, Di Leo S. Providing dignity therapy to patients with advanced cancer: a feasibility study within the setting of a hospital palliative care unit. BMC Palliat Care. 2021 Aug 16;20(1):129. doi: 10.1186/s12904-021-00821-3. PMID 34399737